CLINICAL TRIAL: NCT01616459
Title: Immunogenicity and Safety Study of Two Formulations of GlaxoSmithKline (GSK) Biologicals' Pneumococcal Vaccine (2830929A and 2830930A) When Administered in Healthy Infants
Brief Title: Immunogenicity and Safety of Two Formulations of GSK Biologicals' Pneumococcal Vaccine (2830929A and 2830930A) When Administered in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 116485; 2011-005743-27 (EudraCT Number)
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Infections, Streptococcal
Keywords: Streptococcus pneumoniae; Haemophilus influenzae; Pneumococcal vaccine; Infants; Safety; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Haemophilus Infections | interventions — PHiD-CV vaccine; 13-valent pneumococcal vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 11Pn Group (Experimental): Healthy male or female subjects between, and including 6 to 12 weeks (42-90 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of GSK2830929A, or 11Pn, vaccine at 2, 3 and 4 months of age, followed by a booster dose of the same vaccine at 12-15 months of age, each dose being co-administered with one dose of Infanrix hexa™. The 3 first doses of 11Pn vaccine were administered intramuscularly into the right anterolateral thigh and Infanrix hexa™ was administered intramuscularly into the left anterolateral thigh. The booster dose of 11Pn vaccine was administered intramuscularly into the right deltoid (or thigh if the deltoid muscle size was not adequate) and that of Infanrix hexa™ was administered intramuscularly into the left deltoid (or thigh if the deltoid muscle size was not adequate).
  Interventions: Biological: Pneumococcal conjugate vaccine GSK2830929A; Biological: Infanrix hexa™
- 12Pn Group (Experimental): Healthy male or female subjects between, and including 6 to 12 weeks (42-90 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of GSK2830930A, or 12Pn, vaccine at 2, 3 and 4 months of age, followed by a booster dose of the same vaccine at 12-15 months of age, each dose being co-administered with one dose of Infanrix hexa™. The 3 first doses of 12Pn vaccine were administered intramuscularly into the right anterolateral thigh and Infanrix hexa™ was administered intramuscularly into the left anterolateral thigh. The booster dose of 12Pn vaccine was administered intramuscularly into the right deltoid (or thigh if the deltoid muscle size was not adequate) and that of Infanrix hexa™ was administered intramuscularly into the left deltoid (or thigh if the deltoid muscle size was not adequate).
  Interventions: Biological: Pneumococcal conjugate vaccine GSK2830930A; Biological: Infanrix hexa™
- Synflorix Group (Active Comparator): Healthy male or female subjects between, and including 6 to 12 weeks (42-90 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of Synflorix™ at 2, 3 and 4 months of age, followed by a booster dose of the same vaccine at 12-15 months of age, each dose being co-administered with one dose of Infanrix hexa™. The 3 first doses of Synflorix™ were administered intramuscularly into the right anterolateral thigh and Infanrix hexa™ was administered intramuscularly into the left anterolateral thigh. The booster dose of Synflorix™ was administered intramuscularly into the right deltoid (or thigh if the deltoid muscle size was not adequate) and that of Infanrix hexa™ was administered intramuscularly into the left deltoid (or thigh if the deltoid muscle size was not adequate).
  Interventions: Biological: Synflorix™; Biological: Infanrix hexa™
- Prevnar13 Group (Active Comparator): Healthy male or female subjects between, and including 6 to 12 weeks (42-90 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of Prevnar13™ vaccine at 2, 3 and 4 months of age, followed by a booster dose of the same vaccine at 12-15 months of age, each dose being co-administered with one dose of Infanrix hexa™. The 3 first doses of Prevnar13™ were administered intramuscularly into the right anterolateral thigh and Infanrix hexa™ was administered intramuscularly into the left anterolateral thigh. The booster dose of Prevnar13™ was administered intramuscularly into the right deltoid (or thigh if the deltoid muscle size was not adequate) and that of Infanrix hexa™ was administered intramuscularly into the left deltoid (or thigh if the deltoid muscle size was not adequate ).
  Interventions: Biological: Prevnar 13™; Biological: Infanrix hexa™

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine GSK2830929A — Intramuscular injection
  Arms: 11Pn Group
Biological: Pneumococcal conjugate vaccine GSK2830930A — Intramuscular injection
  Arms: 12Pn Group
Biological: Synflorix™ — Intramuscular injection
  Arms: Synflorix Group
Biological: Prevnar 13™ — Intramuscular injection
  Arms: Prevnar13 Group
Biological: Infanrix hexa™ — Intramuscular injection

SUMMARY:
The purpose of this study is to assess the immunogenicity, reactogenicity and safety of two formulations of GSK Biologicals' pneumococcal vaccine (2830929A and 2830930A) administered as 3-dose primary vaccination during the first 6 months of life followed by a booster dose in the second year of life. To comply with the routine infant immunisation program, the licensed GSK Biologicals DTPa-HBV-IPV/Hib (Infanrix hexa) vaccine will be co-administered in infants with the pneumococcal study vaccines.

DETAILED DESCRIPTION:
The purpose of this study is to assess the immunogenicity of the two formulations of GSK Biologicals' pneumococcal vaccine 2830929A (11-valent vaccine or 11Pn vaccine) and 2830930A (12-valent vaccine or 12Pn vaccine), when administered as 3-dose primary vaccination during the first 6 months of life followed by a booster dose in the second year of life, when compared to immune responses to the licensed vaccines Synflorix™ and Prevnar 13™, and to assess the reactogenicity and safety of these two same investigational formulations when administered according to this schedule. To comply with the routine infant immunisation program, the licensed GSK Biologicals DTPa-HBV-IPV/Hib (Infanrix hexa™) vaccine will be co-administered in infants with the pneumococcal study vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LARs) can and will comply with the requirements of the protocol.
* A male or female between, and including 6 to 12 weeks (42-90 days) of age at the time of the first vaccination. In addition, the first pneumococcal and DTPa-HBV-IPV/Hib vaccination should be given in accordance with the official national recommendations for the immunisation schedule of infants.
* Written informed consent obtained from the parents/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of at least 36 weeks.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/administration of a vaccine containing diphtheria toxoid, tetanus toxoid (except MenC-TT in Spain) or CRM197 and not foreseen by the study protocol during any time of the study period, or of any other vaccines not foreseen by the protocol in the period starting from 30 days before each dose and ending 30 days after each dose of vaccine(s), with the following exceptions:

  * Licensed influenza vaccines are always allowed, even if concomitantly administered with the study vaccines.
  * Licensed rotavirus vaccines are allowed if administered at least 7 days before or after each dose of study of vaccines.
  * Licensed MenC-TT vaccine is allowed in Spain and should be concomitantly administered with the study vaccine at around 2, 4 and 12-15 months of age.
  * In case an emergency mass vaccination for an unforeseen public health threat (e.g. a pandemic) is organised by the public health authorities, outside the routine immunization program, that vaccine can be administered at any time during the study period provided it is licensed and used according to its Summary of Product Characteristics or Prescribing Information and according to the local governmental recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product .
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness, including Kawasaki's syndrome.
* History of any neurological disorders or seizures, including conditions such as hypotensive-hyporesponsive episodes, encephalopathy and any convulsions (afebrile and febrile).
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during study period.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, H. influenzae type b.
* Previous vaccination against S. pneumoniae.
* History of or intercurrent diphtheria, tetanus, pertussis, hepatitis B, polio, H. influenzae type b disease.
* Any medical condition which might interfere with the assessment of the study objectives in the opinion of the investigator.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 953 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2013-04-25 (Actual); Study Completion 2014-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- Czechia (13):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Domažlice
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kladno
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Lipník nad Bečvou
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Ostrov
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- Germany (15):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Schwäbisch Hall, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Berchtesgaden, Bavaria
  - GSK Investigational Site, Kirchheim, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Olching, Bavaria
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Kleve-Materborn, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Wanzleben, Saxony-Anhalt
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Poland (7):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Oleśnica
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Trzebnica
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (6):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Carmona Martinez A, Prymula R, Miranda Valdivieso M, Otero Reigada MDC, Merino Arribas JM, Brzostek J, Szenborn L, Ruzkova R, Horn MR, Jackowska T, Centeno-Malfaz F, Traskine M, Dobbelaere K, Borys D. Immunogenicity and safety of 11- and 12-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccines (11vPHiD-CV, 12vPHiD-CV) in infants: Results from a phase II, randomised, multicentre study. Vaccine. 2019 Jan 3;37(1):176-186. doi: 10.1016/j.vaccine.2018.07.023. Epub 2018 Jul 24. PMID 30054160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 953 subjects were enrolled in the study, among whom 951 received at least one dose of study vaccine, while 2 were allocated a subject number but did not receive any study vaccine dose.
Pre-assignment Details: Study vaccines were administered as a 3-dose primary vaccination in healthy infants between 6-12 weeks (42-90 days) of age at the time of the first vaccination (Primary Phase), and then as an additional booster dose when subjects reached 12-15 months of age (Booster Phase).
Groups:
- Prevnar13 Group: Healthy male or female subjects between, and including 6 to 12 weeks (42-90 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of Prevnar13™ vaccine at 2, 3 and 4 months of age, followed by a booster dose of the same vaccine at 12-15 months of age, each dose being co-administered with one dose of Infanrix hexa™. The 3 first doses of Prevnar13™ were administered intramuscularly into the right anterolateral thigh and Infanrix hexa™ was administered intramuscularly into the left anterolateral thigh. The booster dose of Prevnar13™ was administered intramuscularly into the right deltoid (or thigh if the deltoid muscle size was not adequate) and that of Infanrix hexa™ was administered intramuscularly into the left deltoid (or thigh if the deltoid muscle size was not adequate).
Period: Overall Study
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Started | 240 | 240 | 230 | 241
Completed | 236 | 223 | 220 | 233
Not Completed | 4 | 17 | 10 | 8
Not completed — Adverse Event | 1 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 11 | 3 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 4 | 4 | 4
Not completed — Other reason | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group | Total
Number analyzed (Participants) | 240 | 240 | 230 | 241 | 951
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (1.49) | 8.7 (1.61) | 8.7 (1.62) | 8.6 (1.54) | 8.6 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 120 | 113 | 121 | 467
  Male | 127 | 120 | 117 | 120 | 484

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations Against Pneumococcal Serotypes During the Primary Phase of the Study
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F-Inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. Primary outcome results correspond to antibody concentrations for all serotypes presented at the exception of those for the antibodies against the cross-reactive pneumococcal serotype 3 (ANTI-3).
Time Frame: At study Month 3, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity of the Primary Phase which included all evaluable subjects for whom data concerning primary immunogenicity outcome measures were available for antibodies against at least one vaccine antigen component after primary vaccination against pneumococcal diseases.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 223 | 214 | 210 | 219
µg/mL
  ANTI-1: number analyzed (Participants) | 222 | 214 | 210 | 218
  ANTI-1 | 1.54 [1.37 to 1.74] | 1.59 [1.41 to 1.79] | 1.37 [1.21 to 1.54] | 2.18 [1.97 to 2.42]
  ANTI-3: number analyzed (Participants) | 221 | 214 | 209 | 218
  ANTI-3 | 0.06 [0.05 to 0.06] | 0.06 [0.05 to 0.07] | 0.05 [0.05 to 0.06] | 2.27 [2.06 to 2.49]
  ANTI-4: number analyzed (Participants) | 222 | 214 | 210 | 218
  ANTI-4 | 1.78 [1.56 to 2.02] | 1.99 [1.73 to 2.28] | 1.68 [1.47 to 1.93] | 2.83 [2.60 to 3.09]
  ANTI-5: number analyzed (Participants) | 222 | 214 | 209 | 218
  ANTI-5 | 2.48 [2.24 to 2.74] | 2.37 [2.13 to 2.64] | 2.19 [1.97 to 2.44] | 2.81 [2.52 to 3.13]
  ANTI-6A: number analyzed (Participants) | 222 | 214 | 208 | 218
  ANTI-6A | 0.14 [0.12 to 0.17] | 1.12 [0.93 to 1.34] | 0.12 [0.10 to 0.14] | 2.05 [1.81 to 2.32]
  ANTI-6B: number analyzed (Participants) | 222 | 214 | 210 | 218
  ANTI-6B | 0.51 [0.42 to 0.61] | 0.58 [0.48 to 0.69] | 0.48 [0.40 to 0.58] | 0.49 [0.42 to 0.58]
  ANTI-7F | 2.30 [2.10 to 2.52] | 2.44 [2.18 to 2.72] | 2.20 [1.97 to 2.47] | 3.16 [2.91 to 3.43]
  ANTI-9V: number analyzed (Participants) | 222 | 214 | 210 | 218
  ANTI-9V | 1.57 [1.40 to 1.76] | 1.77 [1.58 to 1.97] | 1.42 [1.27 to 1.59] | 2.27 [2.05 to 2.51]
  ANTI-14: number analyzed (Participants) | 222 | 214 | 210 | 218
  ANTI-14 | 4.19 [3.72 to 4.71] | 4.45 [3.95 to 5.00] | 4.21 [3.72 to 4.77] | 4.20 [3.68 to 4.80]
  ANTI-18C: number analyzed (Participants) | 222 | 214 | 210 | 219
  ANTI-18C | 2.84 [2.45 to 3.28] | 2.56 [2.21 to 2.96] | 2.56 [2.19 to 2.98] | 3.17 [2.87 to 3.51]
  ANTI-19A: number analyzed (Participants) | 222 | 214 | 209 | 219
  ANTI-19A | 1.63 [1.43 to 1.86] | 1.18 [1.03 to 1.36] | 0.18 [0.15 to 0.22] | 2.67 [2.39 to 3.00]
  ANTI-19F: number analyzed (Participants) | 223 | 214 | 210 | 218
  ANTI-19F | 3.65 [3.20 to 4.16] | 3.31 [2.91 to 3.76] | 3.68 [3.15 to 4.30] | 3.07 [2.83 to 3.34]
  ANTI-23F: number analyzed (Participants) | 222 | 214 | 210 | 218
  ANTI-23F | 0.62 [0.52 to 0.73] | 0.69 [0.57 to 0.83] | 0.72 [0.61 to 0.86] | 1.59 [1.38 to 1.84]
Statistical Analysis 1: Comparison: 11Pn Group vs Synflorix Group; ANTI-1 serotype test :to demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC =1.51 in the 11Pn Group and N= 203 and Adjusted GMC= 1.36 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.90, 95.9% CI 2-sided [0.75 to 1.07]
Statistical Analysis 2: Comparison: 11Pn Group vs Synflorix Group; ANTI-4 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC =1.77 in the 11Pn Group and N= 203 and Adjusted GMC= 1.66 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.94, 95.9% CI 2-sided [0.77 to 1.14]
Statistical Analysis 3: Comparison: 11Pn Group vs Synflorix Group; ANTI-5 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC = 2.46 in the 11Pn Group and N= 201 and Adjusted GMC= 2.16 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.88, 95.9% CI 2-sided [0.75 to 1.03]
Statistical Analysis 4: Comparison: 11Pn Group vs Synflorix Group; ANTI-6B serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC =0.51 in the 11Pn Group and N= 200 and Adjusted GMC= 0.47 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.93, 95.9% CI 2-sided [0.71 to 1.23]
Statistical Analysis 5: Comparison: 11Pn Group vs Synflorix Group; ANTI-7F serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=219 and Adjusted GMC =2.30 in the 11Pn Group and N= 202 and Adjusted GMC= 2.17 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.94, 95.9% CI 2-sided [0.81 to 1.10]
Statistical Analysis 6: Comparison: 11Pn Group vs Synflorix Group; ANTI-9V serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC =1.56 in the 11Pn Group and N= 200 and Adjusted GMC= 1.40 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.89, 95.9% CI 2-sided [0.76 to 1.06]
Statistical Analysis 7: Comparison: 11Pn Group vs Synflorix Group; ANTI-14 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC = 4.22 in the 11Pn Group and N= 201 and Adjusted GMC= 4.06 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.96, 95.9% CI 2-sided [0.81 to 1.15]
Statistical Analysis 8: Comparison: 11Pn Group vs Synflorix Group; ANTI-18C serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC =2.81 in the 11Pn Group and N= 201 and Adjusted GMC= 2.57 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 0.92, 95.9% CI 2-sided [0.74 to 1.14]
Statistical Analysis 9: Comparison: 11Pn Group vs Synflorix Group; ANTI-19F serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC = 3.70 in the 11Pn Group and N= 202 and Adjusted GMC= 3.68 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 1.0, 95.9% CI 2-sided [0.81 to 1.23]
Statistical Analysis 10: Comparison: 11Pn Group vs Synflorix Group; ANTI-23F serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=218 and Adjusted GMC = 0.62 in the 11Pn Group and N= 199 and Adjusted GMC= 0.71 for the Synflorix Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 1.15, 95.9% CI 2-sided [0.89 to 1.48]
Statistical Analysis 11: Comparison: 11Pn Group vs Prevnar13 Group; ANTI-19A serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 9 out of 11 vaccine serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.9% CI of the ELISA GMC ratios (Prevnar13/11Pn) and (Synflorix/11Pn) groups < a limit of 2-fold for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — GMCs ratio and its CI were calculated using an ANCOVA model on the logarithm-transformed concentrations/titres, including the vaccine group as fixed effect and the pre-vaccination concentration as regressor. The GMCs were used to calculate the Adjusted GMCs (N=217 and Adjusted GMC =1.61 in the 11Pn Group and N= 206 and Adjusted GMC= 2.75 for the Prevnar13 Group) which in turn were used to calculate the Adjusted GMC ratio with 95.9% confidence interval; Adjusted GMCs ratio = 1.71, 95.9% CI 2-sided [1.44 to 2.03]
Statistical Analysis 12: Comparison: 12Pn Group vs Synflorix Group; ANTI-1 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=207 and Adj. GMC =1.58 in 12Pn Group and N= 203 and Adj. GMC= 1.35 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.86, 95.8% CI [0.72 to 1.02]
Statistical Analysis 13: Comparison: 12Pn Group vs Synflorix Group; ANTI-4 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=208 and Adj. GMC =1.94 in 12Pn Group and N= 203 and Adj. GMC= 1.66 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.86, 95.8% CI [0.70 to 1.05]
Statistical Analysis 14: Comparison: 12Pn Group vs Synflorix Group; ANTI-5 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=208 and Adj. GMC =2.37 in 12Pn Group and N= 201 and Adj. GMC= 2.16 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.91, 95.8% CI 2-sided [0.78 to 1.07]
Statistical Analysis 15: Comparison: 12Pn Group vs Synflorix Group; ANTI-6B serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=208 and Adj. GMC =0.56 in 12Pn Group and N= 200 and Adj. GMC= 0.47 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.84, 95.8% CI [0.64 to 1.11]
Statistical Analysis 16: Comparison: 12Pn Group vs Synflorix Group; ANTI-7F serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=211 and Adj. GMC =2.42 in 12Pn Group and N= 202 and Adj. GMC= 2.17 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.90, 95.8% CI 2-sided [0.76 to 1.06]
Statistical Analysis 17: Comparison: 12Pn Group vs Synflorix Group; ANTI-9V serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=208 and Adj. GMC =1.78 in 12Pn Group and N= 200 and Adj. GMC= 1.40 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.79, 95.8% CI 2-sided [0.67 to 0.93]
Statistical Analysis 18: Comparison: 12Pn Group vs Synflorix Group; ANTI-14 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=209 and Adj. GMC =4.48 in 12Pn Group and N= 201 and Adj. GMC= 4.10 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 0.91, 95.8% CI 2-sided [0.77 to 1.09]
Statistical Analysis 19: Comparison: 12Pn Group vs Synflorix Group; ANTI-18C serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=209 and Adj. GMC =2.55 in 12Pn Group and N= 201 and Adj. GMC= 2.57 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 1.01, 95.8% CI 2-sided [0.81 to 1.26]
Statistical Analysis 20: Comparison: 12Pn Group vs Synflorix Group; ANTI-19F serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=211 and Adj. GMC =3.29 in 12Pn Group and N= 202 and Adj. GMC= 3.67 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 1.12, 95.8% CI 2-sided [0.90 to 1.38]
Statistical Analysis 21: Comparison: 12Pn Group vs Synflorix Group; ANTI-23F serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=208 and Adj. GMC =0.68 in 12Pn Group and N= 199 and Adj. GMC= 0.71 for Synflorix Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 1.05, 95.8% CI 2-sided [0.81 to 1.37]
Statistical Analysis 22: Comparison: 12Pn Group vs Prevnar13 Group; ANTI-6A serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A&19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=210 and Adj. GMC =1.09 in 12Pn Group and N= 214 and Adj. GMC= 2.07 for Prevnar13 Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 1.90, 95.8% CI 2-sided [1.51 to 2.39]
Statistical Analysis 23: Comparison: 12Pn Group vs Prevnar13 Group; ANTI-19A serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™ 1 month post-dose 3 was non-inferior for at least 10 out of 12 vaccine serotypes to Prevnar13 (for 6A&19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of Enzyme-linked immunosorbent assay (ELISA) GMCs. Criteria: UL of the 2-sided 95.8 CI of the ELISA GMC ratios (Prevnar13/12Pn) and (Synflorix/12Pn) groups < a limit of 2-fold for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 12-valent formulation objectives to be assessed sequentially after demonstration for 11-valent formulation. GMCs ratio and its CI obtained using ANCOVA model on logarithm-transformed concentrations, including vaccine group as fixed effect and pre-vaccination concentration as regressor. GMCs were used to calculate Adjusted GMCs (N=208 and Adj. GMC =1.19 in 12Pn Group and N= 206 and Adj. GMC= 2.76 for Prevnar13 Group) which in turn were used to calculate Adjusted GMC ratio with 95.8% CI; Adjusted GMCs ratio = 2.32, 95.8% CI 2-sided [1.94 to 2.77]

2. Primary Outcome: Percentage (%) of Subjects (Synflorix and 11Pn Groups) With Antibody Concentration ≥ 0.2 μg/mL for Pneumococcal Serotypes
Description: N = number of subjects with post primary vaccination results available. % = percentage of subjects with ELISA pneumococcal antibody concentrations ≥ 0.2 μg/mL. Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (ANTI-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F). Antibody concentrations were measured by 22F-Inhibition enzyme-linked immunosorbent assay (ELISA).
Time Frame: 1 month post-dose 3 (primary phase)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity of the Primary Phase which included all evaluable subjects for whom data concerning primary immunogenicity outcome measures were available for antibodies against at least one vaccine antigen component after primary vaccination against pneumococcal diseases.
Measure: Number; unit: Percentage of participants
Arm/Group | 11Pn Group | Synflorix Group
Number analyzed (Participants) | 223 | 210
Percentage of participants
  ANTI-1: number analyzed (Participants) | 222 | 210
  ANTI-1 | 99.5 | 98.6
  ANTI-4: number analyzed (Participants) | 222 | 210
  ANTI-4 | 97.7 | 96.7
  ANTI-5: number analyzed (Participants) | 222 | 209
  ANTI-5 | 100 | 99.5
  ANTI-6B: number analyzed (Participants) | 222 | 210
  ANTI-6B | 77.5 | 75.2
  ANTI-7F | 99.6 | 99.5
  ANTI-9V: number analyzed (Participants) | 222 | 210
  ANTI-9V | 98.6 | 99.0
  ANTI-14: number analyzed (Participants) | 222 | 210
  ANTI-14 | 99.5 | 100
  ANTI-18C: number analyzed (Participants) | 222 | 210
  ANTI-18C | 99.1 | 98.1
  ANTI-19F | 100 | 97.6
  ANTI-23F: number analyzed (Participants) | 222 | 210
  ANTI-23F | 81.1 | 83.8
Statistical Analysis 1: Comparison: 11Pn Group vs Synflorix Group; ANTI-1 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 2-sided 95.9 % Confidence Interval (CI) adjusted 1-sided (alpha = 2.05 %) of the difference between groups in terms of percentage of subjects. Confidence Interval (CI) for difference in proportion: Proc StatXact was used to derive the standardized asymptotic CI for the group difference in proportions [Newcombe, 1998]. The standardized asymptotic method used within GSK Biologicals is method 6; Difference in percentage = -0.98, 95.9% CI 2-sided [-3.89 to 1.36]
Statistical Analysis 2: Comparison: 11Pn Group vs Synflorix Group; ANTI-4 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — 2-sided 95.9% Confidence Interval (CI) adjusted 1-sided (alpha = 2.05 %) of the difference between groups in terms of percentage of subjects. Confidence Interval (CI) for difference in proportion: Proc StatXact was used to derive the standardized asymptotic CI for the group difference in proportions [Newcombe, 1998]. The standardized asymptotic method used within GSK Biologicals is method 6; Difference in percentage = -1.08, 95.9% CI 2-sided [-4.94 to 2.45]
Statistical Analysis 3: Comparison: 11Pn Group vs Synflorix Group; ANTI-5 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = -0.48, 95.9% CI 2-sided [-2.82 to 1.38]
Statistical Analysis 4: Comparison: 11Pn Group vs Synflorix Group; ANTI-6B serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = -2.24, 95.9% CI 2-sided [-10.65 to 6.13]
Statistical Analysis 5: Comparison: 11Pn Group vs Synflorix Group; ANTI-7F serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = -0.03, 95.9% CI 2-sided [-2.39 to 2.21]
Statistical Analysis 6: Comparison: 11Pn Group vs Synflorix Group; ANTI-9V serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = 0.40, 95.9% CI 2-sided [-2.36 to 3.22]
Statistical Analysis 7: Comparison: 11Pn Group vs Synflorix Group; ANTI-14 serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = 0.45, 95.9% CI 2-sided [-1.51 to 2.66]
Statistical Analysis 8: Comparison: 11Pn Group vs Synflorix Group; ANTI-18C serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = -1.00, 95.9% CI 2-sided [-4.18 to 1.70]
Statistical Analysis 9: Comparison: 11Pn Group vs Synflorix Group; ANTI-19F serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = -2.38, 95.9% CI 2-sided [-5.64 to -0.52]
Statistical Analysis 10: Comparison: 11Pn Group vs Synflorix Group; ANTI-23F serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = 2.73, 95.9% CI 2-sided [-4.84 to 10.25]

3. Primary Outcome: Percentage (%) of Subjects (Prevnar13 and 11Pn Groups) With Antibody Concentration ≥ 0.2 μg/mL for Anti-19A Pneumococcal Serotype
Description: N = number of subjects with post primary vaccination results available. % = percentage of subjects with ELISA pneumococcal antibody concentrations ≥ 0.2 μg/mL. Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotype 19A (ANTI-19A). Antibody concentrations were measured by 22F-Inhibition enzyme-linked immunosorbent assay (ELISA).
Time Frame: 1 month post-dose 3 (primary phase)
Population: The analysis was performed on the ATP cohort for immunogenicity of the Primary Phase which included all evaluable subjects for whom data concerning primary immunogenicity outcome measures were available for antibodies against at least one vaccine antigen component after primary vaccination against pneumococcal diseases.
Measure: Number; unit: Percentage of participants
Groups:
- Prevnar13 Group: Healthy male or female subjects between, and including 6 to 12 weeks (42-90 days) of age at the time of first vaccination, received a 3-dose primary vaccination course of Prevnar13™ vaccine at 2, 3 and 4 months of age, followed by a booster dose of the same vaccine at 12-15 months of age, each dose being co-administered with one dose of Infanrix hexa™. The first 3 doses of Prevnar13™ were administered intramuscularly into the right anterolateral thigh and Infanrix hexa™ was administered intramuscularly into the left anterolateral thigh. The booster dose of Prevnar13™ was administered intramuscularly into the right deltoid (or thigh if the deltoid muscle size was not adequate) and that of Infanrix hexa™ was administered intramuscularly into the left deltoid (or thigh if the deltoid muscle size was not adequate).
Arm/Group | 11Pn Group | Prevnar13 Group
Number analyzed (Participants) | 222 | 219
Percentage of participants | 98.6 | 99.5
Statistical Analysis 1: Comparison: 11Pn Group vs Prevnar13 Group; ANTI-19A serotype test: To demonstrate that 11Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 9 out of 11 serotypes to Prevnar13 (for 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.9 % CI of the difference between (Prevnar13 minus 11Pn) and (Synflorix minus 11Pn) groups < 10 % for at least 9 out of 11 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in percentage = 0.89, 95.9% CI 2-sided [-1.46 to 3.66]

4. Primary Outcome: Percentage (%) of Subjects (Synflorix and 12Pn Groups) With Antibody Concentration ≥ 0.2 μg/mL for Pneumococcal Serotypes
Description: as for outcome 2
Time Frame: 1 month post-dose 3 (primary phase)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | 12Pn Group | Synflorix Group
Number analyzed (Participants) | 214 | 210
Percentage of participants
  ANTI-1 | 99.1 | 98.6
  ANTI-4 | 96.7 | 96.7
  ANTI-5: number analyzed (Participants) | 214 | 209
  ANTI-5 | 99.5 | 99.5
  ANTI-6B | 79.9 | 75.2
  ANTI-7F | 99.1 | 99.5
  ANTI-9V | 99.1 | 99.0
  ANTI-14 | 100 | 100
  ANTI-18C | 98.6 | 98.1
  ANTI-19F | 98.6 | 97.6
  ANTI-23F | 81.3 | 83.8
Statistical Analysis 1: Comparison: 12Pn Group vs Synflorix Group; ANTI-1 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — Objectives for 12-valent formulation were to be assessed sequentially after demonstration of objectives for 11-valent formulation. 2-sided 95.8% Confidence Interval (CI) adjusted 1-sided (alpha =2.08%) of the difference between groups in terms of percentage of subjects. CI for difference in proportion: Proc StatXact was used to derive the standardized asymptotic CI for the group difference in proportions [Newcombe,1998]. The standardized asymptotic method used within GSK Biologicals is method 6; Difference in percentage = -0.49, 95.8% CI 2-sided [-3.44 to 2.22]
Statistical Analysis 2: Comparison: 12Pn Group vs Synflorix Group; ANTI-4 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = -0.06, 95.8% CI 2-sided [-4.03 to 3.86]
Statistical Analysis 3: Comparison: 12Pn Group vs Synflorix Group; ANTI-5 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = -0.01, 95.8% CI 2-sided [-2.37 to 2.30]
Statistical Analysis 4: Comparison: 12Pn Group vs Synflorix Group; ANTI-6B serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = -4.67, 95.8% CI 2-sided [-12.94 to 3.60]
Statistical Analysis 5: Comparison: 12Pn Group vs Synflorix Group; ANTI-7F serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = 0.46, 95.8% CI 2-sided [-1.93 to 3.06]
Statistical Analysis 6: Comparison: 12Pn Group vs Synflorix Group; ANTI-9V serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = -0.02, 95.8% CI 2-sided [-2.72 to 2.64]
Statistical Analysis 7: Comparison: 12Pn Group vs Synflorix Group; ANTI-14 serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = 0.00, 95.8% CI 2-sided [-1.94 to 1.90]
Statistical Analysis 8: Comparison: 12Pn Group vs Synflorix Group; ANTI-18C serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = -0.50, 95.8% CI 2-sided [-3.72 to 2.52]
Statistical Analysis 9: Comparison: 12Pn Group vs Synflorix Group; ANTI-19F serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = -0.98, 95.8% CI 2-sided [-4.38 to 2.10]
Statistical Analysis 10: Comparison: 12Pn Group vs Synflorix Group; ANTI-23F serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A and 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups < 10 % for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = 2.50, 95.8% CI 2-sided [-5.07 to 10.06]

5. Primary Outcome: Percentage (%) of Subjects (Prevnar13 and 12Pn Groups) With Antibody Concentration ≥ 0.2 μg/mL for Anti-6A and 19A Pneumococcal Serotypes
Description: N = number of subjects with post primary vaccination results available. % = percentage of subjects with ELISA pneumococcal antibody concentrations ≥ 0.2 μg/mL. Antibodies assessed for this outcome measure were those against the vaccine pneumococcal serotype 6A and 19A (ANTI-6A and 19A). Antibody concentrations were measured by 22F-Inhibition enzyme-linked immunosorbent assay (ELISA).
Time Frame: 1 month post-dose 3 (primary phase)
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | 12Pn Group | Prevnar13 Group
Number analyzed (Participants) | 214 | 219
Percentage of participants
  ANTI-6A: number analyzed (Participants) | 214 | 218
  ANTI-6A | 88.3 | 99.5
  ANTI-19A | 95.8 | 99.5
Statistical Analysis 1: Comparison: 12Pn Group vs Prevnar13 Group; ANTI-6A serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups <10% for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = 11.22, 95.8% CI 2-sided [7.22 to 16.49]
Statistical Analysis 2: Comparison: 12Pn Group vs Prevnar13 Group; ANTI-19A serotype test: To demonstrate that 12Pn co-administered with Infanrix hexa™1 month post-dose 3 was non-inferior for at least 10 out of 12 serotypes to Prevnar13 (for 6A & 19A) or Synflorix™ (for 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F) in terms of % of subjects with antibody concentrations ≥ 0.2 μg/mL. Criteria: UL of 2-sided 95.8 % CI of the difference between (Prevnar13 minus 12Pn) and (Synflorix minus 12Pn) groups <10% for at least 10 out of 12 vaccine pneumococcal serotypes; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in percentage = 3.75, 95.8% CI 2-sided [1.03 to 7.57]

6. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes During the Booster Phase of the Study
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -3, -4, -5, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F-Inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. Analysis of concentrations of antibodies against the cross-reactive pneumococcal serotype 6C (ANTI-6C) will not be performed due to unavailability of a specific qualified assay.
Time Frame: At study Month 10 (M10) and Month 11 (M11), e.g.: prior to and at one month post booster vaccination with pneumococcal vaccine
Population: The analysis was performed on the ATP cohort for immunogenicity of the Booster Phase which included all evaluable subjects for whom data concerning booster immunogenicity outcome measures were available for antibodies against at least one vaccine antigen component before or after booster vaccination against pneumococcal diseases.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 216 | 206 | 203 | 210
µg/mL
  ANTI-1 (M10): number analyzed (Participants) | 216 | 206 | 202 | 210
  ANTI-1 (M10) | 0.26 [0.24 to 0.30] | 0.26 [0.24 to 0.30] | 0.26 [0.23 to 0.29] | 0.44 [0.40 to 0.48]
  ANTI-1 (M11): number analyzed (Participants) | 214 | 203 | 201 | 209
  ANTI-1 (M11) | 2.49 [2.21 to 2.82] | 2.18 [1.94 to 2.46] | 2.25 [2.01 to 2.53] | 3.84 [3.50 to 4.22]
  ANTI-3 (M10): number analyzed (Participants) | 214 | 204 | 199 | 208
  ANTI-3 (M10) | 0.06 [0.05 to 0.07] | 0.06 [0.05 to 0.06] | 0.06 [0.05 to 0.07] | 0.25 [0.22 to 0.29]
  ANTI-3 (M11): number analyzed (Participants) | 210 | 202 | 197 | 209
  ANTI-3 (M11) | 0.07 [0.06 to 0.08] | 0.07 [0.06 to 0.08] | 0.07 [0.06 to 0.09] | 1.68 [1.53 to 1.85]
  ANTI-4 (M10): number analyzed (Participants) | 213 | 203 | 203 | 210
  ANTI-4 (M10) | 0.49 [0.44 to 0.54] | 0.48 [0.43 to 0.54] | 0.50 [0.45 to 0.56] | 0.41 [0.37 to 0.46]
  ANTI-4 (M11): number analyzed (Participants) | 214 | 203 | 202 | 209
  ANTI-4 (M11) | 3.89 [3.49 to 4.34] | 4.18 [3.77 to 4.63] | 4.06 [3.70 to 4.45] | 3.86 [3.43 to 4.35]
  ANTI-5 (M10): number analyzed (Participants) | 213 | 202 | 199 | 208
  ANTI-5 (M10) | 0.51 [0.46 to 0.57] | 0.51 [0.45 to 0.57] | 0.48 [0.43 to 0.53] | 0.77 [0.69 to 0.85]
  ANTI-5 (M11): number analyzed (Participants) | 215 | 203 | 202 | 209
  ANTI-5 (M11) | 3.23 [2.88 to 3.64] | 3.31 [2.98 to 3.68] | 3.05 [2.75 to 3.38] | 6.84 [6.12 to 7.66]
  ANTI-6B (M10): number analyzed (Participants) | 213 | 202 | 199 | 209
  ANTI-6B (M10) | 0.57 [0.49 to 0.65] | 0.64 [0.56 to 0.74] | 0.59 [0.51 to 0.69] | 0.22 [0.19 to 0.25]
  ANTI-6B (M11): number analyzed (Participants) | 214 | 205 | 203 | 209
  ANTI-6B (M11) | 2.66 [2.34 to 3.03] | 4.09 [3.60 to 4.66] | 2.53 [2.24 to 2.86] | 3.80 [3.34 to 4.33]
  ANTI-7F (M10): number analyzed (Participants) | 213 | 203 | 200 | 207
  ANTI-7F (M10) | 1.04 [0.94 to 1.16] | 0.99 [0.89 to 1.10] | 0.94 [0.84 to 1.05] | 1.21 [1.11 to 1.32]
  ANTI-7F (M11): number analyzed (Participants) | 214 | 203 | 201 | 209
  ANTI-7F (M11) | 4.88 [4.40 to 5.40] | 4.57 [4.14 to 5.04] | 4.31 [3.91 to 4.75] | 6.34 [5.80 to 6.95]
  ANTI-9V (M10): number analyzed (Participants) | 213 | 202 | 198 | 207
  ANTI-9V (M10) | 0.76 [0.68 to 0.85] | 0.77 [0.69 to 0.87] | 0.70 [0.63 to 0.77] | 0.53 [0.48 to 0.58]
  ANTI-9V (M11): number analyzed (Participants) | 214 | 203 | 202 | 209
  ANTI-9V (M11) | 4.14 [3.70 to 4.62] | 4.36 [3.93 to 4.84] | 3.68 [3.32 to 4.09] | 5.83 [5.26 to 6.46]
  ANTI-14 (M10): number analyzed (Participants) | 214 | 204 | 201 | 209
  ANTI-14 (M10) | 1.30 [1.11 to 1.53] | 1.45 [1.28 to 1.64] | 1.12 [0.97 to 1.30] | 1.66 [1.44 to 1.93]
  ANTI-14 (M11): number analyzed (Participants) | 213 | 203 | 201 | 209
  ANTI-14 (M11) | 6.17 [5.45 to 6.98] | 6.52 [5.80 to 7.33] | 5.75 [5.07 to 6.51] | 10.05 [8.97 to 11.25]
  ANTI-18C (M10): number analyzed (Participants) | 212 | 200 | 195 | 207
  ANTI-18C (M10) | 0.76 [0.67 to 0.86] | 0.68 [0.60 to 0.77] | 0.74 [0.65 to 0.84] | 0.59 [0.54 to 0.65]
  ANTI-18C (M11): number analyzed (Participants) | 213 | 203 | 201 | 209
  ANTI-18C (M11) | 7.65 [6.79 to 8.61] | 7.20 [6.39 to 8.11] | 8.00 [7.06 to 9.06] | 6.01 [5.45 to 6.63]
  ANTI-19A (M10): number analyzed (Participants) | 212 | 199 | 197 | 208
  ANTI-19A (M10) | 0.46 [0.39 to 0.54] | 0.36 [0.31 to 0.42] | 0.18 [0.15 to 0.21] | 0.42 [0.35 to 0.49]
  ANTI-19A (M11): number analyzed (Participants) | 214 | 203 | 201 | 209
  ANTI-19A (M11) | 5.35 [4.67 to 6.13] | 4.46 [3.83 to 5.20] | 1.11 [0.91 to 1.35] | 7.06 [6.25 to 7.98]
  ANTI-19F (M10): number analyzed (Participants) | 212 | 199 | 196 | 207
  ANTI-19F (M10) | 1.11 [0.97 to 1.28] | 1.11 [0.96 to 1.29] | 1.10 [0.95 to 1.29] | 0.50 [0.44 to 0.57]
  ANTI-19F (M11): number analyzed (Participants) | 213 | 203 | 203 | 209
  ANTI-19F (M11) | 8.67 [7.72 to 9.73] | 8.50 [7.55 to 9.59] | 8.22 [7.40 to 9.13] | 6.40 [5.77 to 7.11]
  ANTI-23F (M10): number analyzed (Participants) | 214 | 205 | 198 | 208
  ANTI-23F (M10) | 0.51 [0.44 to 0.58] | 0.54 [0.47 to 0.62] | 0.49 [0.43 to 0.56] | 0.34 [0.29 to 0.39]
  ANTI-23F (M11): number analyzed (Participants) | 214 | 203 | 201 | 209
  ANTI-23F (M11) | 3.09 [2.73 to 3.49] | 3.31 [2.93 to 3.73] | 2.98 [2.65 to 3.35] | 6.49 [5.69 to 7.39]

7. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes During the Primary Phase of the Study
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine/cross-reactive pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19F and 23F (OPA-1, -3, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19F and -23F). The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8. Testing for opsonophagocytic activity against the cross-reactive pneumococcal serotype 6C will not be performed due to unavailability of a specific qualified assay.
Time Frame: At study Month 3, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 105 | 105 | 99 | 105
Titers
  OPA-1: number analyzed (Participants) | 105 | 105 | 98 | 105
  OPA-1 | 13.2 [9.6 to 18.2] | 15.6 [11.4 to 21.1] | 13.6 [9.9 to 18.6] | 26.4 [19.3 to 36.0]
  OPA-3: number analyzed (Participants) | 101 | 100 | 94 | 100
  OPA-3 | 4.8 [4.2 to 5.5] | 5.2 [4.4 to 6.0] | 5.0 [4.3 to 5.7] | 97.2 [81.6 to 116.0]
  OPA-4: number analyzed (Participants) | 103 | 105 | 99 | 104
  OPA-4 | 527.3 [401.5 to 692.4] | 609.0 [492.8 to 752.5] | 616.7 [503.2 to 756.0] | 540.1 [444.7 to 656.1]
  OPA-5: number analyzed (Participants) | 102 | 104 | 98 | 105
  OPA-5 | 43.0 [32.6 to 56.9] | 46.7 [36.8 to 59.3] | 40.5 [30.4 to 54.0] | 57.2 [44.3 to 74.0]
  OPA-6A: number analyzed (Participants) | 100 | 103 | 94 | 103
  OPA-6A | 37.4 [22.9 to 60.9] | 1292.6 [940.3 to 1777.0] | 36.5 [22.6 to 59.0] | 2832.0 [2212.8 to 3624.4]
  OPA-6B: number analyzed (Participants) | 101 | 104 | 96 | 103
  OPA-6B | 478.3 [345.2 to 662.7] | 603.2 [436.9 to 832.8] | 622.6 [444.2 to 872.7] | 742.3 [533.9 to 1031.8]
  OPA-7F: number analyzed (Participants) | 104 | 103 | 98 | 104
  OPA-7F | 3515.0 [2787.1 to 4433.0] | 4472.3 [3463.6 to 5774.9] | 3424.1 [2631.9 to 4454.8] | 9737.9 [7540.5 to 12575.8]
  OPA-9V: number analyzed (Participants) | 105 | 105 | 98 | 104
  OPA-9V | 1212.9 [953.6 to 1542.6] | 1629.0 [1293.0 to 2052.4] | 1469.9 [1178.3 to 1833.6] | 1614.5 [1283.9 to 2030.2]
  OPA-14: number analyzed (Participants) | 105 | 104 | 97 | 103
  OPA-14 | 1000.8 [743.1 to 1347.9] | 1699.1 [1313.8 to 2197.3] | 1417.4 [1059.6 to 1896.0] | 2034.4 [1513.4 to 2734.8]
  OPA-18C: number analyzed (Participants) | 105 | 102 | 98 | 102
  OPA-18C | 100.9 [67.7 to 150.4] | 131.5 [86.9 to 198.8] | 72.0 [47.0 to 110.4] | 145.7 [102.6 to 206.8]
  OPA-19F: number analyzed (Participants) | 102 | 102 | 96 | 103
  OPA-19F | 144.2 [101.8 to 204.3] | 201.4 [147.2 to 275.4] | 210.4 [143.6 to 308.2] | 66.0 [49.8 to 87.5]
  OPA-23F: number analyzed (Participants) | 104 | 104 | 98 | 104
  OPA-23F | 989.6 [652.9 to 1499.8] | 1377.9 [951.5 to 1995.3] | 1097.3 [742.1 to 1622.4] | 5136.4 [3829.2 to 6889.8]

8. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes During the Booster Phase of the Study
Description: as for outcome 7
Time Frame: At study Month 11, e.g.: at one month post booster vaccination with pneumococcal vaccine
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 99 | 97 | 96 | 101
Titers
  OPA-1 | 192.4 [129.0 to 287.1] | 192.4 [133.3 to 277.5] | 216.8 [148.3 to 316.9] | 207.6 [145.8 to 295.6]
  OPA-3: number analyzed (Participants) | 93 | 89 | 85 | 96
  OPA-3 | 9.7 [7.5 to 12.7] | 10.5 [8.0 to 13.7] | 10.9 [7.6 to 15.5] | 317.2 [275.4 to 365.4]
  OPA-4: number analyzed (Participants) | 96 | 96 | 95 | 100
  OPA-4 | 1455.3 [1208.9 to 1751.9] | 1650.5 [1360.9 to 2001.9] | 1550.5 [1230.2 to 1954.1] | 1972.2 [1586.3 to 2451.9]
  OPA-5: number analyzed (Participants) | 99 | 96 | 96 | 100
  OPA-5 | 134.5 [100.3 to 180.4] | 133.3 [105.2 to 168.8] | 133.4 [100.5 to 177.1] | 269.9 [216.2 to 337.0]
  OPA-6A: number analyzed (Participants) | 95 | 93 | 92 | 98
  OPA-6A | 116.8 [67.9 to 201.0] | 3436.7 [2716.0 to 4348.5] | 146.4 [87.6 to 244.6] | 5200.7 [4134.9 to 6541.3]
  OPA-6B: number analyzed (Participants) | 98 | 96 | 95 | 100
  OPA-6B | 681.4 [520.3 to 892.5] | 1246.4 [963.1 to 1613.0] | 694.6 [546.5 to 882.6] | 1727.9 [1406.2 to 2123.4]
  OPA-7F: number analyzed (Participants) | 96 | 96 | 96 | 97
  OPA-7F | 8362.9 [6977.1 to 10023.9] | 7516.4 [6223.0 to 9078.7] | 7880.8 [6408.6 to 9691.3] | 16592.6 [13909.7 to 19792.9]
  OPA-9V: number analyzed (Participants) | 99 | 97 | 93 | 96
  OPA-9V | 3406.9 [2758.2 to 4208.1] | 3616.1 [2838.1 to 4607.5] | 3260.6 [2620.1 to 4057.6] | 8470.4 [6692.4 to 10720.8]
  OPA-14: number analyzed (Participants) | 99 | 96 | 94 | 100
  OPA-14 | 2038.4 [1594.3 to 2606.2] | 2519.9 [1960.2 to 3239.6] | 2285.1 [1845.9 to 2828.9] | 2772.6 [2218.6 to 3464.9]
  OPA-18C: number analyzed (Participants) | 97 | 95 | 93 | 97
  OPA-18C | 914.8 [621.8 to 1345.9] | 781.2 [536.3 to 1137.8] | 912.0 [605.4 to 1374.1] | 610.7 [421.3 to 885.1]
  OPA-19F: number analyzed (Participants) | 95 | 96 | 96 | 98
  OPA-19F | 523.9 [382.9 to 716.8] | 565.3 [406.4 to 786.6] | 759.6 [554.3 to 1040.8] | 438.0 [312.7 to 613.7]
  OPA-23F: number analyzed (Participants) | 97 | 96 | 95 | 97
  OPA-23F | 2562.9 [2016.3 to 3257.6] | 2923.6 [2248.9 to 3800.9] | 2600.0 [1896.8 to 3563.9] | 24350.4 [18303.2 to 32395.5]

9. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) During the Primary Phase of the Study
Description: Anti-PD antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The cut-off of the assay was an anti-PD antibody concentration higher than or equal to (≥) 100 EL.U/mL.
Time Frame: At study Month 3, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 112 | 106 | 103 | 106
EL.U/mL | 1430.1 [1194.2 to 1712.7] | 1194.2 [1017.7 to 1401.3] | 1344.8 [1116.4 to 1619.9] | 64.4 [57.7 to 71.9]

10. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) During the Booster Phase of the Study
Description: as for outcome 9
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 108 | 102 | 101 | 106
EL.U/mL
  Anti-PD (M10) | 445.9 [365.0 to 544.7] | 447.6 [363.4 to 551.2] | 460.0 [376.2 to 562.4] | 70.9 [61.8 to 81.3]
  Anti-PD (M11): number analyzed (Participants) | 108 | 100 | 101 | 104
  Anti-PD (M11) | 1866.0 [1535.7 to 2267.4] | 1835.5 [1511.5 to 2229.0] | 2128.4 [1777.1 to 2549.2] | 77.8 [67.1 to 90.1]

11. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms During the Primary Phase
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm).
Time Frame: Within the 4-day (Days 0-3) post-vaccination period following each primary dose (D).
Population: The analysis was performed on the Total Vaccinated cohort for the Primary Phase, which included all subjects who received at least one of the 3 vaccine doses priming against pneumococcal diseases, with analysis done solely on subjects for whom post-vaccination results about solicited symptoms were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 240 | 236 | 228 | 238
Participants
  Any Pain, post D1 | 104 | 105 | 94 | 85
  Grade 3 Pain, post D1 | 16 | 5 | 12 | 6
  Any Redness, post D1 | 82 | 90 | 72 | 75
  Grade 3 Redness, post D1 | 0 | 0 | 1 | 0
  Any Swelling, post D1 | 51 | 57 | 46 | 47
  Grade 3 Swelling, post D1 | 1 | 4 | 7 | 1
  Any Pain, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Pain, post D2 | 89 | 100 | 88 | 90
  Grade 3 Pain, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Pain, post D2 | 12 | 12 | 10 | 6
  Any Redness, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Redness, post D2 | 86 | 95 | 78 | 79
  Grade 3 Redness, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Redness, post D2 | 2 | 1 | 1 | 1
  Any Swelling, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Swelling, post D2 | 61 | 72 | 54 | 49
  Grade 3 Swelling, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Swelling, post D2 | 2 | 3 | 5 | 2
  Any Pain, post D3: number analyzed (Participants) | 238 | 229 | 226 | 234
  Any Pain, post D3 | 76 | 75 | 76 | 75
  Grade 3 Pain, post D3: number analyzed (Participants) | 238 | 229 | 226 | 234
  Grade 3 Pain, post D3 | 4 | 4 | 6 | 3
  Any Redness, post D3: number analyzed (Participants) | 238 | 229 | 226 | 234
  Any Redness, post D3 | 93 | 85 | 91 | 85
  Grade 3 Redness, post D3: number analyzed (Participants) | 238 | 229 | 226 | 234
  Grade 3 Redness, post D3 | 3 | 2 | 2 | 1
  Any Swelling, post D3: number analyzed (Participants) | 238 | 229 | 226 | 234
  Any Swelling, post D3 | 72 | 76 | 58 | 61
  Grade 3 Swelling, post D3: number analyzed (Participants) | 238 | 229 | 226 | 234
  Grade 3 Swelling, post D3 | 2 | 5 | 2 | 3

12. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms During the Booster Phase of the Study
Description: as for outcome 11
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort for the Booster Phase, which included all subjects who received the booster dose against pneumococcal diseases, with analysis done solely on subjects for whom post-vaccination results about solicited symptoms were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 235 | 224 | 219 | 231
Participants
  Any Pain | 112 | 123 | 119 | 110
  Grade 3 Pain | 13 | 16 | 18 | 8
  Any Redness | 109 | 117 | 108 | 107
  Grade 3 Redness | 5 | 10 | 7 | 5
  Any Swelling | 84 | 88 | 89 | 85
  Grade 3 Swelling | 8 | 7 | 5 | 7

13. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination, During the Primary Phase of the Study
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness (Irr./Fuss.), Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than [≥] 38.0 degrees Celsius [°C]),. Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Rectal temperature higher than (>) 40.0°C.
Time Frame: Within the 4-day (Days 0-3) post-vaccination period following each primary dose (D).
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 240 | 236 | 227 | 238
Participants
  Any Drowsiness, post D1 | 148 | 144 | 129 | 129
  Grade 3 Drowsiness, post D1 | 7 | 6 | 10 | 10
  Related Drowsiness, post D1 | 124 | 104 | 95 | 103
  Any Irr./Fuss., post D1 | 151 | 156 | 134 | 138
  Grade 3 Irr./Fuss., post D1 | 16 | 15 | 17 | 10
  Related Irr./Fuss., post D1 | 119 | 122 | 98 | 103
  Any Loss Appet., post D1 | 85 | 89 | 81 | 73
  Grade 3 Loss Appet., post D1 | 2 | 2 | 3 | 2
  Related Loss Appet., post D1 | 59 | 65 | 56 | 57
  Any Fever, post D1 | 108 | 104 | 107 | 87
  Grade 3 Fever, post D1 | 0 | 0 | 0 | 0
  Related Fever, post D1 | 94 | 91 | 92 | 76
  Any Drowsiness, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Drowsiness, post D2 | 125 | 115 | 105 | 111
  Grade 3 Drowsiness, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Drowsiness, post D2 | 6 | 7 | 6 | 8
  Related Drowsiness, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Related Drowsiness, post D2 | 96 | 89 | 81 | 97
  Any Irr./Fuss., post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Irr./Fuss., post D2 | 151 | 151 | 141 | 128
  Grade 3 Irr./Fuss., post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Irr./Fuss., post D2 | 18 | 12 | 17 | 10
  Related Irr./Fuss., post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Related Irr./Fuss., post D2 | 123 | 113 | 114 | 106
  Any Loss Appet., post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Loss Appet., post D2 | 69 | 78 | 71 | 72
  Grade 3 Loss Appet., post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Loss Appet., post D2 | 2 | 3 | 1 | 3
  Related Loss Appet., post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Related Loss Appet., post D2 | 52 | 58 | 48 | 56
  Any Fever, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Any Fever, post D2 | 97 | 84 | 90 | 90
  Grade 3 Fever, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Grade 3 Fever, post D2 | 0 | 0 | 0 | 0
  Related Fever, post D2: number analyzed (Participants) | 239 | 232 | 227 | 234
  Related Fever, post D2 | 87 | 75 | 82 | 82
  Any Drowsiness, post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Any Drowsiness, post D3 | 99 | 92 | 88 | 87
  Grade 3 Drowsiness, post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Grade 3 Drowsiness, post D3 | 4 | 2 | 3 | 5
  Related Drowsiness, post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Related Drowsiness, post D3 | 80 | 67 | 70 | 71
  Any Irr./Fuss., post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Any Irr./Fuss., post D3 | 117 | 123 | 118 | 112
  Grade 3 Irr./Fuss., post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Grade 3 Irr./Fuss., post D3 | 6 | 7 | 8 | 7
  Related Irr./Fuss., post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Related Irr./Fuss., post D3 | 95 | 92 | 96 | 87
  Any Loss Appet., post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Any Loss Appet., post D3 | 63 | 62 | 67 | 54
  Grade 3 Loss Appet., post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Grade 3 Loss Appet., post D3 | 0 | 3 | 3 | 5
  Related Loss Appet., post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Related Loss Appet., post D3 | 49 | 42 | 54 | 41
  Any Fever, post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Any Fever, post D3 | 51 | 53 | 61 | 58
  Grade 3 Fever, post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Grade 3 Fever, post D3 | 0 | 0 | 0 | 0
  Related Fever, post D3: number analyzed (Participants) | 238 | 229 | 227 | 234
  Related Fever, post D3 | 50 | 51 | 56 | 49

14. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination, During the Booster Phase of the Study
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness (Irr./Fuss.), Loss of appetite (Loss Appet.) and Fever (rectal temperature higher than [≥] 38.0 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irr./Fuss. = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = Rectal temperature higher than (>) 40.0°C.
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 235 | 224 | 219 | 231
Participants
  Any Drowsiness | 109 | 100 | 84 | 96
  Grade 3 Drowsiness | 9 | 6 | 4 | 2
  Related Drowsiness | 93 | 79 | 68 | 81
  Any Irr./Fuss. | 140 | 136 | 137 | 129
  Grade 3 Irr./Fuss. | 14 | 14 | 12 | 9
  Related Irr./Fuss. | 107 | 117 | 109 | 107
  Any Loss Appet. | 80 | 85 | 83 | 61
  Grade 3 Loss Appet. | 6 | 3 | 9 | 7
  Related Loss Appet. | 66 | 64 | 65 | 45
  Any Fever. | 80 | 72 | 68 | 75
  Grade 3 Fever | 2 | 0 | 1 | 0
  Related Fever | 72 | 66 | 60 | 67

15. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) During the Primary Phase of the Study
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination.
Time Frame: Within the 31-day (Days 0-30) period post primary vaccination, across doses
Population: The analysis was performed on the Total Vaccinated cohort for the Primary Phase, which included all subjects who received at least one of the 3 vaccine doses priming against pneumococcal diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 240 | 240 | 230 | 241
Participants | 110 | 108 | 123 | 124

16. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) During the Booster Phase of the Study
Description: as for outcome 15
Time Frame: Within the 31-day (Days 0-30) period post booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort for the Booster Phase, which included all subjects who received the booster dose against pneumococcal diseases.
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 237 | 226 | 222 | 234
Participants | 69 | 68 | 74 | 53

17. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)During the Primary Phase of the Study
Description: A SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalisation, as per the medical or scientific judgement of the physician. Any = Occurrence of a SAE, regardless of relationship to vaccination.
Time Frame: From Month 0 to Month 3
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 240 | 240 | 230 | 241
Participants | 12 | 11 | 17 | 12

18. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) During the Entire Duration of the Study
Description: A SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalisation, as per the medical or scientific judgement of the the physician. Any = Occurrence of a SAE, regardless of relationship to vaccination.
Time Frame: From Day 0 to Month 11
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 240 | 240 | 230 | 241
Participants | 29 | 26 | 38 | 24

19. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotype 6A During the Booster Phase of the Study
Description: Antibodies assessed for this outcome measure was that against the cross-reactive pneumococcal serotype 6A (ANTI-6A). Antibody concentrations were measured by 22F-Inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL.
Time Frame: as for outcome 6
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity of the Booster Phase which included all evaluable subjects for whom data concerning booster immunogenicity outcome measures were available for antibodies against at least one vaccine antigen component before or after booster vaccination against pneumococcal diseases.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 212 | 203 | 200 | 209
µg/mL
  ANTI-6A (M10): number analyzed (Participants) | 211 | 196 | 194 | 205
  ANTI-6A (M10) | 0.23 [0.19 to 0.27] | 0.89 [0.78 to 1.01] | 0.22 [0.18 to 0.26] | 0.64 [0.56 to 0.73]
  ANTI-6A (M11) | 1.07 [0.90 to 1.27] | 7.94 [6.99 to 9.02] | 0.91 [0.76 to 1.09] | 9.31 [8.41 to 10.30]

20. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes 19A During the Primary Phase of the Study
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine/cross-reactive pneumococcal serotypes 19A (OPA-19A). The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) serotype-specific Lower Limit of Quantification (143).
Time Frame: At study Month 3, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 87 | 88 | 76 | 92
Titers | 1813.0 [1524.4 to 2156.1] | 1523.9 [1215.3 to 1910.9] | 759.6 [559.2 to 1032.0] | 2056.6 [1748.9 to 2418.4]

21. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes 19A During the Booster Phase of the Study
Description: as for outcome 20
Time Frame: At study Month 11, e. g. at one month post-Booster vaccination with pneumococcal vaccine
Population: as for outcome 19
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 74 | 67 | 69 | 75
Titers | 4866.4 [4184.6 to 5659.4] | 3896.4 [3263.2 to 4652.4] | 2191.0 [1720.0 to 2791.0] | 5720.1 [4883.9 to 6699.4]

22. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotype 6C During the Primary Phase of the Study.
Description: No analysis was performed on Enzyme-Linked ImmunoSorbent Assay (ELISA) testing for antibody concentrations against vaccine serotype 6C as no specific qualified/validated assay was available.
Time Frame: At study Month 3, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: The analysis was to be performed on the According-to-Protocol cohort for immunogenicity of the Primary Phase. But no analysis was performed on Enzyme-Linked ImmunoSorbent Assay (ELISA) testing for antibody concentrations against vaccine serotype 6C as no specific qualified/validated assay was available
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

23. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotype 6C During the Booster Phase of the Study.
Description: as for outcome 22
Time Frame: as for outcome 6
Population: The analysis was to be performed on the According-to-Protocol cohort for immunogenicity of the Booster Phase but no analysis was performed on Enzyme-Linked ImmunoSorbent Assay (ELISA) testing for antibody concentrations against vaccine serotype 6C as no specific qualified/validated assay was available.
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

24. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes 6C During the Primary Phase of the Study
Description: No analysis was performed on opsonophagocytic activity for antibody titers against vaccine serotype 6C as no specific qualified/validated assay was available.
Time Frame: At study Month 3, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: The analysis was to be performed on the According-to-Protocol cohort for immunogenicity of the Primary Phase but no analysis was performed on opsonophagocytic activity for antibody titers against vaccine serotype 6C as no specific qualified/validated assay was available.
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes 6C During the Booster Phase of the Study
Description: as for outcome 24
Time Frame: At study Month 11, e. g. at one month post-Booster vaccination with pneumococcal vaccine
Population: The analysis was to be performed on the According-to-Protocol cohort for immunogenicity of the Booster Phase but no analysis was performed on opsonophagocytic activity for antibody titers against vaccine serotype 6C as no specific qualified/validated assay was available.
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 4 days post-primary and post-booster vaccination. Unsolicited AEs: during 31 days post-primary and post-booster vaccination. SAEs: during the whole study period (from Day 0 to Month 11).
Description: Analysis of AEs and SAEs was performed on all subjects who received at least one primary vaccination dose or at least the booster vaccination. Analysis of solicited symptoms was performed on subjects who received at least one primary vaccination or at least the booster vaccination and for whom results were available.
Arm/Group | 11Pn Group | 12Pn Group | Synflorix Group | Prevnar13 Group
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/240 | 0/230 | 0/241
Serious Adverse Events (participants affected / at risk) | 29/240 | 26/240 | 38/230 | 24/241
Other Adverse Events (participants affected / at risk) | 234/240 | 229/240 | 221/230 | 235/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 11Pn Group (N=240) | 12Pn Group (N=240) | Synflorix Group (N=230) | Prevnar13 Group (N=241)
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Pyrexia (General disorders) | 0 | 4 | 1 | 0 — SAE reported between Day 0 and Month 11
Milk allergy (Immune system disorders) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Bacteraemia (Infections and infestations) | 0 | 1 | 1 | 0 — SAE reported between Day 0 and Month 11
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Bronchiolitis (Infections and infestations) | 5 | 1 | 2 | 3 — SAE reported between Day 0 and Month 11
Bronchitis (Infections and infestations) | 5 | 1 | 7 | 4 — SAE reported between Day 0 and Month 11
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 1 — SAE reported between Day 0 and Month 11
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Gastroenteritis (Infections and infestations) | 2 | 2 | 1 | 2 — SAE reported between Day 0 and Month 11
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1 — SAE reported between Day 0 and Month 11
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 — SAE reported between Day 0 and Month 11
Pertussis (Infections and infestations) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Pneumonia (Infections and infestations) | 3 | 2 | 3 | 1 — SAE reported between Day 0 and Month 11
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 2 | 0 | 1 — SAE reported between Day 0 and Month 11
Pyelonephritis (Infections and infestations) | 0 | 0 | 4 | 0 — SAE reported between Day 0 and Month 11
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1 | 5 | 1 — SAE reported between Day 0 and Month 11
Tracheitis (Infections and infestations) | 1 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 2 — SAE reported between Day 0 and Month 11
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 — SAE reported between Day 0 and Month 11
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 — SAE reported between Day 0 and Month 11
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 — SAE reported between Day 0 and Month 11
Hypotonic-hyporesponsive episode (Nervous system disorders) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Febrile convulsion (Nervous system disorders) | 0 | 1 | 2 | 1 — SAE reported between Day 0 and Month 11
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 2 | 1 — SAE reported between Day 0 and Month 11
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 — SAE reported between Day 0 and Month 11
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Impetigo (Infections and infestations) | 0 | 0 | 1 | 1 — SAE reported between Day 0 and Month 11
Otitis media (Infections and infestations) | 0 | 0 | 2 | 0 — SAE reported between Day 0 and Month 11
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 — SAE reported between Day 0 and Month 11
Adenoiditis (Infections and infestations) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Escherichia pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Gastroenteritis adenovirus (Infections and infestations) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Intervertebral discitis (Infections and infestations) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Otitis media acute (Infections and infestations) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 — SAE reported between Day 0 and Month 11
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Pyomyositis (Infections and infestations) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Retinoblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 — SAE reported between Day 0 and Month 11
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 — SAE reported between Day 0 and Month 11
Viral tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 — SAE reported between Day 0 and Month 11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 11Pn Group (N=240) | 12Pn Group (N=240) | Synflorix Group (N=230) | Prevnar13 Group (N=241)
Pain (General disorders) | 140 | 141/236 | 134/228 | 126/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Redness (General disorders) | 132 | 144/236 | 130/228 | 134/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Swelling (General disorders) | 108 | 117/236 | 91/228 | 93/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Drowsiness (General disorders) | 185 | 178/236 | 162/228 | 168/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Irritability/Fussiness (General disorders) | 202 | 203/236 | 185/228 | 186/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Loss of appetite (General disorders) | 124 | 132/236 | 125/228 | 125/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Fever (rectal temperature ≥ 38°C) (General disorders) | 153 | 144/236 | 148/228 | 143/238 — Symptom reported during the 4-day post-primary vaccination periods , across doses
Upper respiratory tract infection (Infections and infestations) | 38 | 39 | 49 | 28 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Rhinitis (Infections and infestations) | 18 | 15 | 12 | 16 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Bronchiolitis (Infections and infestations) | 12 | 10 | 13 | 11 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Bronchitis (Infections and infestations) | 10 | 7 | 18 | 16 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Nasopharyngitis (Infections and infestations) | 10 | 14 | 8 | 11 — Unsolicited AE reported during the 31-day post-primary vaccination periods, across doses
Pain (General disorders) | 112/235 | 123/224 | 119/219 | 110/231 — Symptom reported during the 4-day post-booster vaccination period
Redness (General disorders) | 109/235 | 117/224 | 108/219 | 107/231 — Symptom reported during the 4-day post-booster vaccination period
Swelling (General disorders) | 84/235 | 88/224 | 89/219 | 85/231 — Symptom reported during the 4-day post-booster vaccination period
Drowsiness (General disorders) | 109/235 | 100/224 | 84/219 | 96/231 — Symptom reported during the 4-day post-booster vaccination period
Irritability/Fusiness (General disorders) | 140/235 | 136/224 | 137/219 | 129/231 — Symptom reported during the 4-day post-booster vaccination period
Loss of appetite (General disorders) | 80/235 | 85/224 | 83/219 | 61/231 — Symptom reported during the 4-day post-booster vaccination period
Fever (rectal temperature ≥ 38°C) (General disorders) | 80/235 | 72/224 | 68/219 | 75/231 — Symptom reported during the 4-day post-booster vaccination period
Upper respiratory tract infection (Infections and infestations) | 11/237 | 16/226 | 20/222 | 13/234 — Unsolicited AE reported during the 31-day post-booster vaccination period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.